CLINICAL TRIAL: NCT05678712
Title: Improved Glycemic Control in Diabetic Patients in Hemodialysis Using Continuous Glucose Monitoring (CGM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Steno Diabetes Center Nordjylland (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Peter Vestergaard, MD, professor, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N-20210070
Record Dates: First submitted 2022-03-04; First posted 2023-01-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hemodialysis; Type1diabetes; Type2Diabetes
Keywords: Diabetes; Heamodialysis; CGM; Glycemic control; Algorithm
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention): After a two weeks "run-in" baseline period (blinded CGM) some of the participants (1:1) were randomly assigned to six weeks of standard treatment, i.e. self monitoring of blood glucose (the last two weeks with blinded CGM → 2 weeks "wash-out" (baseline for next period) (blinded CGM) → six weeks with non-blinded CGM with data available for the patient himself/herself and dialysis staff
- Intervention (access to CGM data) (Experimental): After a two weeks "run-in" baseline period (blinded CGM) some of the participants (1:1) were randomly assigned to six weeks with non-blinded CGM with data available for the patient himself/herself and dialysis staff → 2 weeks "wash-out" (baseline for next period) (blinded CGM) → Six weeks of standard treatment, i.e. self monitoring of blood glucose (the last two weeks with blinded CGM
  Interventions: Device: Access to CGM data (Dexcom G6)

INTERVENTIONS:
Device: Access to CGM data (Dexcom G6) — Acces to CGM data (not blinded CGM)
  Arms: Intervention (access to CGM data)

SUMMARY:
The 16-week trial is an open-label cross-over trial which includes heamodialysis patients with T2D and T1D on insulin therapy. During one period, patients carry a non-blinded CGM. In the other period they follow standard procedures (the last two weeks with a blinded CGM). The patients and the dialysis staff can use the CGM measures to regulate insulin and food intake during the non-blinded weeks. The research group will collect the CGM-data during the trial.

DETAILED DESCRIPTION:
Background: Managing diabetes is often problematic in haemodialysis (HD) patients. Low blood glucose is especially common during treatment. Typically, the patient's blood sugar is only measured during treatment if considered relevant. Otherwise, HbA1c is used to control diabetes - a method associated with uncertain in HD patients. An alternative or supplement to the current management of diabetes could be CGM which enables closer observation and management of the diabetes disease. Despite the possibilities of using CGM, there are still few studies in the field which examine the importance of CGM data in relation to the management of diabetes in HD patients.

Aims: To investigate whether the use of CGM data can prevent low blood sugar levels during HD and examins whether the use of CGM data can improve the management of diabetes in HD patients. Furthermore, it is found relevant to investigate if CGM data, selected blood test responses, treatment data, personal data and information about medicines can be used to predict low blood sugar during HD using an algorithm. Thus, the study also aims to develop and validate such an algorithm.

Setting: The trial will be conducted at two dialysis wards (Aalborg and Hjørring) at Aalborg University Hospital.

Subjects: Heamodialysis patients with T1D and T2D on insulin therapy.

Study design: The 16-week trial is an open-label cross-over trial. During one period, patients carry a non-blinded CGM. In the other period they follow standard procedures (the last two weeks with a blinded CGM). The patients and the dialysis staff can use the CGM measures to regulate insulin and food intake during the non-blinded weeks. The research group will collect the CGM-data during the trial. The last four weeks include baseline measures (blinded CGM).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Chronically ill heamodialysis patients (heamodialysis or heamodiafiltration - treatment)der modtager HD- eller hæmodiafiltrationsbehandling på dialyseafsnit,--
* Patients at dialysis wards in Aalborg and Hjørring, Aalborg University Hospital (center and home patients)
* T1D or T2D and in treatment with insulin
* Being able to use CGM equipment
* Signed consent

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Terms that, in the opinion of the investigator or subinvestigators, render the participant unfit to conduct the trial, including lack of understanding of the trial or lack of physical or cognitive ability to participate
* Patients undergoing peritoneal dialysis (PD) or heamofiltration dialysis (HF)
* Acute HD treatment
* Gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
time below range (CGM) | 6 weeks of treatment in each of the two treatment periods
  Change in time below range (CGM) (< 3.0 mmol/L)

SECONDARY OUTCOMES:
Time in range (CGM) | 6 weeks of treatment in each of the two treatment periods
  Change in time in range (CGM) (3,9-10,0 mmol/L)
Time in borderline low range (CGM) | 6 weeks of treatment in each of the two treatment periods
  Change in CGM time in low range(3.0 mmol/L ≤ glucose < 3.9 mmol/L)
Time above range (CGM) | 6 weeks of treatment in each of the two treatment periods
  Change in CGM time above range (>10 mmol/L)
Time above range (CGM) (high) | 6 weeks of treatment in each of the two treatment periods
  Change in CGM time above range (>13,9 mmol/L)
Concentration of HbA1c | 6 weeks of treatment in each of the two treatment periods
  Change in HbA1c
Glucose variability | 6 weeks of treatment in each of the two treatment periods
  Glucose variability (variation coefficient or SD)
Sensitivity and specificity of algorithm | Through study completion, an average of one year
  Sensitivity and specificity of algorithm to predict hypoglycemias

OTHER OUTCOMES:
Hypo- and hyperglycemic episodes | 6 weeks of treatment in each of the two treatment periods
  Number of hypo- and hyperglycemic episodes (15 minutes)
Insulin requirements | 6 weeks of treatment in each of the two treatment periods
  Changes in insulin requirements based on detection/memorisation (with help from nurse) of insulin doses and time points
Diabetes-related quality of life | Week 0, week 6, week 8, week 14
  Assessing whether there is a difference between intervention and standard treatment. Measured using the Dawn-2 Impact of Diabetes Questionnaire (DIDP) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sisse Heiden Laursen, PhD, Principal Investigator — Aalborg University; Peter Vestergaard, PhD (and MD), Study Chair — Aalborg University Hospital and Steno Diabetes Center
Locations (1):
- Department of nephrology (dialysis), Aalborg, Denmark